CLINICAL TRIAL: NCT01917058
Title: A Randomized Clinical Trial to Evaluate the Efficacy of Abatacept in Moderate to Severe Alopecia Areata
Brief Title: A Clinical Trial to Evaluate the Efficacy of Abatacept in Moderate to Severe Alopecia Areata
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unfortunately we did not receive funding and therefore were not able to begin the trial.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Julian M. Mackay-Wiggan, Principal Investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAL0950
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Abatacept
MeSH Terms: conditions — Alopecia Areata | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abatacept (Active Comparator)
  Interventions: Drug: Abatacept
- abatacept Subcutaneous vehicle (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Abatacept — This will be a randomized double blind placebo controlled study. Patients will be randomly assigned to abatacept or placebo in a 1:1 ratio based on a computer generated randomization list. The list will be generated prior to study initiation. Based on the randomization list, patients will be assigned to treatment vs. vehicle (provided by BMS) in the order in which they are enrolled. The assignment will be made by study personnel who are not involved in making clinical assessments or evaluations. The patient and the assessing physicians will remain blinded to the treatment assignment for the duration of the study.
  Patients will be treated with abatacept 125mg SC self-administered each week. Treatment will be continued for 6 months to provide adequate time to assess the short-term efficacy and safety of abatacept in patients with alopecia areata. Patients will then be followed for an additional 6 months to assess the timing and incidence of relapse.
  Other Names: Brand Name: ORENCIA
  Arms: abatacept
Drug: placebo
  Arms: abatacept Subcutaneous vehicle

SUMMARY:
The purpose of this study is to determine if receiving sub-cutaneous injections of a medication called abatacept causes regrowth of hair in people with alopecia areata.

Among patients with alopecia areata, patients with worse disease are unlikely to have satisfactory outcomes with current therapies. Our hypothesis is that Abatacept will be effective therapy in moderate to severe alopecia areata by blocking re-activation of a special type of immunecell call a memory T-Cell (CD8+NKG2D+)thereby blocking the inflammatory response underlying alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a common disease of the immune system, known as an "autoimmune" disease. In the disease, the immune system mistaken destroys the hair follicle, causing hair to fall out. Despite many people having this disease, research into its cause and into new, better ways to treat AA has lagged far behind other similar diseases of the immune system. Currently, there are no Federal Drug Administration approved drugs for AA. Abatacept (made by Bristol-Myers Squibb) is a safe intervention known to effectively treat rheumatoid arthritis,another "autoimmune" disease, by fighting inflammation. There are some genetic and chemical similarities between those with active rheumatoid arthritis and AA, suggesting that treatment with the same drug is likely to be effective.

In mice specially designed for testing drugs for the treatment of human alopecia, this medication worked to prevent the disease AA from starting. To test Abatacept, we are going to treat 60 patients with moderate to severe AA for 6 months. To make the study results meaningful, there will be a control or "placebo" group that does not receive the study drug. Patients will be randomly assigned to either receive the real or the inactive medication, and neither the patient nor the doctor will know which it is. The effectiveness of the medication will be measured by changes in hair re-growth as determined by physical exam and photography, as well as by patient and physician scoring. Patients will be followed for another 6 months off of the drug to see if the effects of treatment last and if there is delayed response. Small scalp biopsies and peripheral blood will be taken at the beginning of the study before treatment and then after 4,12 and 24 weeks. The chemical analysis of these skin samples and blood will help us to understand how the disease happens, how the treatment works, and even guide us to better treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Must be between 18 and 75 years of age.
* Must have a diagnosis of moderate to severe AA - defined as the presence of equal to or more than 40% and equal to or less than 95% total scalp hair loss at baseline as measured using the SALT score.
* Duration of hair loss must be between 3 to 12 months.
* There may be no evidence of regrowth present at baseline.
* Subjects may be naïve to treatment or unresponsive to intralesional (IL) steroids or other treatments for AA.
* Must be willing to avoid live vaccines while on the study medication, and within 3 months of its discontinuation.
* Women of childbearing potential must use highly effective methods of birth control [for up to 12 weeks after the last dose of investigational product] to minimize the risk of pregnancy].
* Women of childbearing potential must follow instructions for birth control for the entire duration of the study including a minimum of 90 days after dosing has been completed.
* Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
* Women must not be breastfeeding
* Sexually active fertile men must use highly effective birth control if their partners are women of childbearing potential.
* Men that are sexually active with women of childbearing potential must follow instructions for birth control for the entire duration of the study and a minimum of 90 days after dosing has been completed.

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study drug.
* Women of childbearing potential using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or before administration of abatacept.
* Sexually active fertile men not using effective birth control if their partners are women of childbearing potential.
* Patients with alopecia totalis/universalis
* Patients with a history of or active skin disease on the scalp such as psoriasis or seborrheic dermatitis.
* Patients in whom the diagnosis of alopecia areata is in question.
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma) that in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
* Patients with COPD
* Patients known to be HIV or hepatitis B or C positive.
* Patients with history or evidence of hematopoietic abnormality.
* Patients with history of immunosuppression or history of recurrent serious infections.
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in AA
* Patients taking TNF antagonists or other biological therapy such as anakinra.
* Patients known to be HIV or hepatitis B or C positive.
* Patients with evidence of infection or active/untreated skin cancer.
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.
* Subjects who are impaired, incapacitated, or incapable of completing study-related assessments.
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
* Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ.

Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.

* Subjects who currently abuse drugs or alcohol.
* Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
* Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
* Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
* Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (e.g., chronic pyelonephritis, osteomyelitis, or bronchiectasis).
* Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
* Subjects must not be positive for HIV, Hepatitis B or C.
* Subjects who are positive for hepatitis C antibody
* Subjects who have at any time received treatment with any investigational drug within 28 days
* Any concomitant biologic Disease Modifying Anti-Rheumatic Drugs (DMARDS), such as anakinra.
* Subjects who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.

OTHER EXCLUSION CRITERIA

* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
SALT Score (Severity of Alopecia Tool) | 24 Weeks
  The primary efficacy endpoint of this intention-to-treat trial will be the proportion of responders in the treated compared to the control group after 6 months of treatment, defined as 50% or greater hair re-growth from baseline as assessed by SALT score at week 24. This patient group and relatively strict definition for defining responders were chosen to minimize responses in the "vehicle" arm, in which 8% are expected to achieve this magnitude of hair regrowth spontaneously. To assess the durability of responses, patients who achieve 50% regrowth from baseline during the first 6 months, will continue to be followed for an additional 6 months off treatment or until it is determined that relapse has occurred.

SECONDARY OUTCOMES:
Efficacy | 24 Weeks of Treatment and an additional 6 months off treatment or until determined that relapse has ocurred
  Efficacy will be measured by changes in hair re-growth as a continuous variable as determined by physical exam and Canfield photography, as well as patient and physician global evaluation scores. To assess the durability of responses, patients who achieve 50% regrowth from baseline during the first 6 months, will continue to be followed for an additional 6 months off treatment or until it is determined that relapse has occurred.
Safety | 24 Weeks of Treatment and an additional 6 months off treatment or until determined that relapse has ocurred
  Patient reported outcomes, safety measures, incidence and timing of relapse will be important secondary outcomes.
  Safety will be evaluated as a secondary endpoint using descriptive statistics to summarize the cumulative incidence and types of Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Dept of Dermatology, New York, New York, United States